CLINICAL TRIAL: NCT00556946
Title: Combined Photodynamic and Pulsed Dye Laser Treatment of Port Wine Stains
Acronym: PDT/PDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor of Dermatology and Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20033286
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stains
Keywords: Vascular Malformation
MeSH Terms: conditions — Hemangioma, Capillary; Vascular Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Photodynamic & Pulsed Dye Laser Treatment (Other): Treatment of Port Wine Stains
  Interventions: Drug: Combined Photodynamic & Pulsed Dye Laser Treatment

INTERVENTIONS:
Drug: Combined Photodynamic & Pulsed Dye Laser Treatment — Treatment of Port Wine Stains using Combined Photodynamic and Pulsed Dye Laser

SUMMARY:
This research study was designed to determine the effect on port wine stains (PWS) of liposomal benzoporphyrin derivative monoacid (BPD-MA) termed verteporfin by intravenous (IV) infusion for photodynamic therapy (PDT) or combined PDT and pulsed dye laser (PDL) therapy (PDT + PDL). The standard treatment for PWS is PDL alone. This lightens some PWS but many lesions are not completely removed.

PDT uses a medication and light together to cause injury to a target. The medication is given and then light is directed at the desired area of treatment to achieve an effect. PDT has been used to treat some skin conditions including pre-cancers and skin cancers. Using PDT or PDT immediately followed by PDL therapy may improve PWS lightening. At this time, both PDT and PDT + PDL therapy for treatment of PWS is investigational. The type and amount of medication and light which may be used to treat PWS is not known, and is likely to be different than those used for other PDT treatments.

DETAILED DESCRIPTION:
Procedures will be performed at the Surgery Laser Clinic at the Beckman Laser Institute at the University of California, Irvine.

At an initial visit, a brief history and physical will be performed.

The history will include: 1) previous treatment to my PWS; 2) current medications; 3) history of light sensitivity; 4) risk of pregnancy and use of birth control in a female of child-bearing age.

The physical will include: 1) measurement and evaluation of PWS; 2) measurement of blood pressure, blood cell count, general chemistries (including liver function tests) and ANA, which might indicate an increased sensitivity to light.

On the day of treatment, the same brief physical and history will be repeated. A urine pregnancy test will be performed on females of child-bearing age.

Four circular test sites of PWS will be selected. One test site will receive no treatment. The second test sites will be treated with the pulsed dye laser at standard setting and protective eyeglasses to shield the eyes during the laser treatment.

For two additional test spots, the photodynamic therapy (PDT) verteporfin will be administered intravenously over a 10-minute period. After receiving the verteporfin, the skin and eyes will be sensitive to light for the next 5 days. The light sensitive protection precautions will be instructed.

Optical Doppler Tomography unit (ODT) measurements, similar to shining a flash light to PWS and measuring the light response, which provide information about how blood is flowing through the PWS.

Photographs and light measurements will be taken during follow-up visits on day 1, day 3, and 1, 2, 4, 8 and 12 weeks after the study treatment. At these visits blood may also be drawn to check for blood substances that promote blood vessel formation.

At the end of the study, blood tests will be drawn to assess cell count and general chemistries.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* Have a PWS on an area other than the face
* A negative pregnancy test and non pregnant or nursing

Exclusion Criteria:

* Under 18 years of age
* Have an allergy to verteporfin, porfimer sodium or other porphyrins
* Have a history of porphyria (a disease that can cause sensitivity to light)
* Have had treatment to the PWS test sites in the last 8 weeks
* Have an active uncontrolled infection or other significant disease
* Currently using medications that cause sensitivity to light such as tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics and griseofulvin
* Currently using medications that increase bleeding, including aspirin, coumadin or non-steroidal anti-inflammatory drugs
* Have very dark skin which is sensitive to laser treatment
* Have a positive ANA (lab tests which indicates sensitivity to light)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Medical Clinic,University, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Photodynamic and Pulsed Dye Laser Treatment: Treatment of Port Wine Stains: using Combined Photodynamic and Pulsed Dye Laser.
Period: Overall Study
Arm/Group | Combined Photodynamic and Pulsed Dye Laser Treatment
Started | 17
Completed | 16
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Combined Photodynamic and Pulsed Dye Laser Treatment: Treatment of Port Wine Stains using Combined Photodynamic and Pulsed Dye Laser.
Arm/Group | Combined Photodynamic and Pulsed Dye Laser Treatment
Number analyzed (Participants) | 17
Age, Customized [Number; unit: participants]
  Adult over 18 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Blanching of Port Wine Stain Birthmark
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Treatment of Port Wine Stains: Treatment of Port Wine Stains
  Treatment of Port Wine Stains: Treatment of Port Wine Stains
Arm/Group | Treatment of Port Wine Stains
Number analyzed (Participants) | 16
participants | 16

ADVERSE EVENTS:
Time Frame: Through the study up to 6 weeks
Arm/Group | Treatment of Port Wine Stains
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No